CLINICAL TRIAL: NCT01211236
Title: Maggot Therapy for Wound Debridement: a Randomized Multicentric Double-blind Trial
Brief Title: Maggot Therapy for Wound Debridement
Acronym: MAGGOT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Collaborators: Société de Dermatologie Française (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PHRC04-130
Record Dates: First submitted 2010-09-28; First posted 2010-09-29 (Estimated); Last update posted 2010-09-29 (Estimated); Status verified 2010-09

CONDITIONS: Pressure Ulcers
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Maggot Debridement Therapy (Experimental)
  Interventions: Other: application of wound dressing made of bio-bags (vitapads) containing maggots
- control (Active Comparator)
  Interventions: Other: application of classical hydrogel/alginate wound dressing

INTERVENTIONS:
Other: application of wound dressing made of bio-bags (vitapads) containing maggots
  Arms: Maggot Debridement Therapy
Other: application of classical hydrogel/alginate wound dressing
  Arms: control

SUMMARY:
The main objective of the trial was to study the efficacy of bagged larvae on wound debridement in comparison to classical treatments. The secondary outcome was to assess wound healing, treatment related pain, microbiological modifications, adverse events, comfort of the dressing and duration of wound care. We performed a randomized, double-blind, multicenter, controlled, prospective phase III trial in three referral institutional centers of hospitalized care in Caen, Lisieux and Lyon, France. A total of 120 patients with a non-healing fibrinous wound ≤ 40cm2, less than 2cm-deep, and an ankle-brachial pressure index (ABPI) ≥ 0.8 were included, from March 2005 to December 2008. During two weeks´ hospitalization, patients received either Maggot Debridement Therapy (MDT, changes of bagged larvae twice a week) or classical treatments (mechanical debridement and classical dressings performed three times a week). At discharge, classical dressings were applied and a follow-up visit performed at D30. Main outcome measure was the comparison of the reduction of fibrin percentage on wounds treated with MDT and classical treatments at D15. The percentages of fibrin were measured using a computerized planimetry software package, Canvas (ACD Systems, British Columbia, Canada), which enables the quantification of color surface variations in a wound after manual delimitation (using a mouse) on a series of photographic images.

ELIGIBILITY:
Inclusion Criteria:

* patient between 18 and 90 years old
* patients with a non-healing fibrinous wound ≤ 40cm2 (pressure ulcer or venous ulcers
* pressure ulcers were less than 2cm-deep
* limb wounds were venous ulcers with an ankle-brachial pressure (ABP)≥ 0.8
* signed informed consent

Exclusion Criteria:

* patients pregnant or lactating
* patients with neuropathy
* patients perforant ulcer of the foot
* patients with dementia

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2006-02

PRIMARY OUTCOMES:
Percent of Fibrin changes from day 0 to day 15

SECONDARY OUTCOMES:
Percent of healing changes from day 0 to day 15

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Hospital of Caen, dermatology department, Caen, Calvados
  - Robert Bisson Hospital, Lisieux, Calvados
  - Hopital des armées Desgenettes, Lyon, Rhone

REFERENCES:
- [Derived] Opletalova K, Blaizot X, Mourgeon B, Chene Y, Creveuil C, Combemale P, Laplaud AL, Sohyer-Lebreuilly I, Dompmartin A. Maggot therapy for wound debridement: a randomized multicenter trial. Arch Dermatol. 2012 Apr;148(4):432-8. doi: 10.1001/archdermatol.2011.1895. Epub 2011 Dec 19. PMID 22184720